CLINICAL TRIAL: NCT07116291
Title: Impact of Regular Karate Practice on the Quality of Life and Health Outcomes of Students
Acronym: KARACADEMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC25_0307
Record Dates: First submitted 2025-07-18; First posted 2025-08-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Medical Student

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Karate (Experimental)
  Interventions: Other: Karate
- usual sporting practice except karate (No Intervention)

INTERVENTIONS:
Other: Karate — karate practice
  Arms: Karate

SUMMARY:
A recent study reported that 52% of medical students had an anxiety disorder and 18% had a depressive syndrome. Following this publication, the Inspectorate General of Social Affairs commissioned a report on the quality of life of health students, making it a health priority.

One of the causes of the malaise felt by students could be the stress associated with exams and recent reforms. This malaise could also be due to a drop in self-esteem linked to the environment and atmosphere on certain placement sites. In fact, one of our recent studies suggested that the quality of life of doctors in the clerkship could influence the quality of life of students.

Since self-esteem is an important parameter in a student's understanding of his or her academic career, improving self-esteem could improve academic results and the quality of life of students.

Among the martial arts evaluated, karate has shown promising results in improving concentration and regulating the feelings of child victims of war in particular, as well as the elderly. Karate could therefore be a simple and effective solution for improving the mental health of healthy students, as well as their academic results. As it is a sport considered to be of moderate intensity, particularly through the practice of kat, it can be practised by anyone without contraindication apart from coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* 3rd or 4th year health students at the university of Angers

Exclusion Criteria:

* contraindication to the practice of karate
* students repeating a year or entering the third year after a transfer, insofar as the evolution of their grades in relation to the 2nd year class cannot be ascertained.
* Students who already practise karate regularly cannot be included.
* Students planning to transfer to another faculty during the year of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
evolution of the Short-Form-36 score (SF-36) | 10 months

SECONDARY OUTCOMES:
Evolution of Rosenberg scale score | 10 months
  evolution of self-esteem
evolution of the Pittsburg scale | 10 months
  student sleep quality
ranking students after their exams | 10 months
  Assessment of the evolution of the ranking students in their class according to the ranking of the previous year

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien VENARA, MD-PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- University of ANGERS, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided